CLINICAL TRIAL: NCT02028208
Title: Clinical Evaluation of Metal Panel Allergens: Mercury, Aluminum and Palladium Dose Response Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allerderm (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SP12 2PM2 201
Record Dates: First submitted 2014-01-02; First posted 2014-01-07 (Estimated); Results first posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-04

CONDITIONS: Contact Dermatitis
Keywords: Patch Test; Allergy Testing; Contact Dermatitis; Mercury, Aluminum or Palladium skin allergy
MeSH Terms: conditions — Dermatitis, Contact

STUDY DESIGN:
Intervention Model Description: Biologic
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ammoniated mercury (Experimental): Subjects will be patch tested with 4 experimental doses of ammoniated mercury, 0.013 mg/cm², 0.040 mg/cm², 0.12 mg/cm², and 0.36 mg/cm², a negative control and corresponding reference allergens, 1.0% ammoniated mercury in petrolatum and 0.5% elemental mercury in petrolatum. Patch tests will be worn for 48 hours.
  Interventions: Diagnostic Test: Ammoniated mercury
- Aluminum chloride and aluminum lactate (Experimental): Subjects will be patch tested with 4 experimental doses of aluminum chloride, 0.040 mg/cm², 0.12 mg/cm², 0.36 mg/cm² and 0.72 mg/cm², 4 experimental doses of aluminum lactate 0.047 mg/cm², 0.14 mg/cm², 0.42 mg/cm² and 0.84 mg/cm², a negative control and corresponding reference allergens, 2.0% aluminum chloride in petrolatum and 12.0% aluminum lactate in petrolatum. Patch tests will be worn for 48 hours.
  Interventions: Diagnostic Test: Aluminum chloride and aluminum lactate
- Sodium tetrachloropalladaate (Palladium) (Experimental): Subjects will be patch tested with 5 experimental doses of sodium tetrachloropalladate 0.011 mg/cm², 0.033 mg/cm², 0.10 mg/cm², 0.30 mg/cm² and 0.60 mg/cm², a negative control and corresponding reference allergens, 3.0% sodium tetrachloropalladate in petrolatum and 1.0% palladium chloride 1.0% in petrolatum. Patch tests will be worn for 48 hours.
  Interventions: Diagnostic Test: Sodium tetrachloropalladate

INTERVENTIONS:
Diagnostic Test: Ammoniated mercury — Metal allergen panel containing ascending doses of ammoniated mercury and a negative control.
  Arms: Ammoniated mercury
Diagnostic Test: Aluminum chloride and aluminum lactate — Metal allergen panel containing ascending doses of alumium chloride, aluminum lactate and a negative control.
  Arms: Aluminum chloride and aluminum lactate
Diagnostic Test: Sodium tetrachloropalladate — Metal allergen panel containing ascending doses of sodium tetrachloropalladate and a negative control.
  Arms: Sodium tetrachloropalladaate (Palladium)

SUMMARY:
The purpose of this study is to evaluate the diagnostic performance and safety of ascending doses of mercury, aluminum and palladium metal allergens proposed for inclusion in a metal allergen panel. Optimal dose will be selected based on the lowest dose of each allergen eliciting a positive response in 70-90% of subjects tested.

DETAILED DESCRIPTION:
This is a single-center, double-blind, randomized study to compare the diagnostic performance (primary) and safety (secondary) of ascending doses of mercury, aluminum and palladium in 20 adult subjects who have a clinical history of contact dermatitis and have had a past positive patch test to one of the allergens on this study. Investigators and subjects will be blinded to the exact location of each dose within the allergen panel but will not be blinded to the allergen being tested, nor the range of allergen doses within each panel.

ELIGIBILITY:
Inclusion Criteria:

1.15 years of age or older.

2. History of contact dermatitis.

3. Positive patch results to 1) mercury (elemental), 2) aluminum (aluminum chloride hexahydrate, aluminum hydroxide and/or aluminum lactate) or 3) palladium (sodium tetrachloropalladate and/or palladium chloride) within the past 10 years.

4. Male or non-pregnant non-lactating female. Female subjects must state, at visit one that they are not pregnant, not lactating nor are they intending to become pregnant for the course of the study.

5. Has understood and signed the approved Informed Consent/Assent Form, which is consistent with all institutional, local and national regulations. Assent Form for all minor subjects (ages 15-17) must be signed by the guardian/parent.

Exclusion Criteria:

1. Breastfeeding or pregnant or intending to become pregnant for the course of the study.
2. Topical treatment with corticosteroids or other immunosuppressive agents on or near the test area during the 7 days prior to inclusion in this study.
3. Systemic treatment with corticosteroids (equivalent to > 10 mg prednisone) or other immunosuppressive agents during the 7 days prior to inclusion in this study. Inhaled treatments are permitted.
4. Treatment with ultraviolet (UV) light (including tanning) during the 3 weeks prior to inclusion in this study.
5. Acute dermatitis outbreak or dermatitis on or near the test area on the back.
6. Inability to comply with patch test study requirements including multiple return visits and activity restrictions (e.g., protecting test panels from excess moisture due to showering or vigorous activity).
7. Participation in a clinical trial of an investigational drug, treatment or device other than T.R.U.E. TEST during this study or 3 weeks prior to inclusion in this study.
8. An opinion of the Investigator that deems the potential subject to be non-compliant, unable to return for study visits or complete the study as detailed in the protocol.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-11-04 (Actual); Primary Completion 2016-05-24 (Actual); Study Completion 2016-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Isaksson, MD, Principal Investigator — Skane University Hospital Malmo
Locations (1):
- Skane University Hospital Malmo, Malmo, Sweden

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ammoniated Mercury | Aluminum Chloride and Aluminum Lactate | Sodium Tetrachloropalladaate (Palladium)
Started | 21 | 13 | 22
Completed | 21 | 13 | 21
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ammoniated Mercury | Aluminum Chloride and Aluminum Lactate | Sodium Tetrachloropalladaate (Palladium) | Total
Number analyzed (Participants) | 21 | 13 | 22 | 56
Age, Customized [Count of Participants; unit: Participants] | 21 | 13 | 22 | 56
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 10 | 21 | 47
  Male | 5 | 3 | 1 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Indigenous swede | 6 | 10 | 16 | 32
  Ethnic Sami | 0 | 0 | 0 | 0
  Ethnic Finn | 0 | 1 | 0 | 1
  Other | 15 | 2 | 6 | 23
Region of Enrollment [Number; unit: participants]
  Sweden | 14 | 13 | 22 | 49
  Italy | 7 | 0 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Exhibit Positive Responses to Each Allergen Concentration
Description: Subjects were patch tested with 4 doses of mercury (0.00mg/cm2-neg control, 0.013 mg/cm2-dose 1, 0.040 mg/cm2-dose 2, 0.12 mg/cm2-dose 3 and 0.36 mg/cm2-dose 4) or 0 doses of aluminum (0.00 mg/cm2-neg control, 0.40 mg/cm2 aluminum chloride-dose 1, 0.12 mg/cm2 aluminum chloride-dose 2, 0.36 mg/cm2 aluminum chloride-dose 3 and 0.72 mg/cm2 aluminum chloride-dose 4, 0.047mg/cm2 aluminum lactate-dose 5, 0.14 mg/cm2 aluminum lactate-dose 6, 0.42 mg/cm2 aluminum lactate-dose 7, 0.84 mg/cm2 aluminum lactate-dose 8) or 5 doses of palladium (0.00 mg/cm2-neg control, 0.011 mg/cm2- dose 1, 0.033 mg/cm2- dose 2, 0.10 mg/cm2- dose 3, 0.30 mg/cm2- dose 4 and 0.60 mg/cm2- dose 5)..Skin reactions were assessed at 3, 4 and 21 days following application. A response is considered positive if it is graded 1+, 2+ or 3+during at least one post removal visit. Overall results are based on Investigator determination following the final study visit.
Time Frame: Patch test sites were evaluated at days 3, 7, 10, 14, and 21 days after application. Results are based on Investigator's review of reactions following the day 21 evaluation
Population: Not all subjects were tested with all allergens. Each panel had a different number of ascending doses.
Measure: Count of Participants; unit: Participants
Arm/Group | Ammoniated Mercury | Aluminum Chloride and Aluminum Lactate | Sodium Tetrachloropalladaate (Palladium)
Number analyzed (Participants) | 21 | 13 | 21
Participants
  Negative Control: Number Positive | 4 | 0 | 0
  Negative Control: Number Doubtful | 2 | 2 | 0
  Negative Control: Number Irritant | 0 | 0 | 0
  Negative Control: Number Negative | 15 | 11 | 21
  Dose 1: Number Positive | 10 | 0 | 6
  Dose 1: Number Doubtful | 5 | 1 | 9
  Dose 1: Number Irritant | 0 | 0 | 0
  Dose 1: Number Negative | 6 | 12 | 6
  Dose 2: Number Positive | 16 | 0 | 13
  Dose 2: Number Doubtful | 2 | 1 | 6
  Dose 2: Number Irritant | 1 | 0 | 0
  Dose 2: Number Negative | 2 | 12 | 2
  Dose 3: Number Positive | 14 | 1 | 15
  Dose 3: Number Doubtful | 2 | 3 | 2
  Dose 3: Number Irritant | 0 | 0 | 0
  Dose 3: Number Negative | 5 | 9 | 4
  Dose 4: Number Positive | 15 | 2 | 18
  Dose 4: Number Doubtful | 3 | 6 | 2
  Dose 4: Number Irritant | 0 | 0 | 0
  Dose 4: Number Negative | 3 | 5 | 1
  Dose 5: number analyzed (Participants) | 0 | 13 | 21
  Dose 5: Number Positive |  | 0 | 20
  Dose 5: Number Doubtful |  | 0 | 0
  Dose 5: Number Irritant |  | 0 | 0
  Dose 5: Number Negative |  | 13 | 1
  Dose 6: number analyzed (Participants) | 0 | 13 | 0
  Dose 6: Number Positive |  | 0 |
  Dose 6: Number Doubtful |  | 1 |
  Dose 6: Number Irritant |  | 0 |
  Dose 6: Number Negative |  | 12 |
  Dose 7: number analyzed (Participants) | 0 | 13 | 0
  Dose 7: Number Positive |  | 0 |
  Dose 7: Number Doubtful |  | 3 |
  Dose 7: Number Irritant |  | 0 |
  Dose 7: Number Negative |  | 10 |
  Dose 8: number analyzed (Participants) | 0 | 13 | 0
  Dose 8: Number Positive |  | 1 |
  Dose 8: Number Doubtful |  | 5 |
  Dose 8: Number Irritant |  | 0 |
  Dose 8: Number Negative |  | 7 |
Statistical Analysis 1: Comparison: Ammoniated Mercury; Concordance between Investigational and Reference Allergen presented for allergen doses which met the minimum criteria of 70% with positive reactions; Test type: Other — Concordance between 0.40 mg/cm2 mercury and 1.0% ammoniated mercury in petrolatum; Kappa statistic = 0.38, 95% CI 2-sided [0.08 to 0.67]
Statistical Analysis 2: Comparison: Ammoniated Mercury; [analysis description as in outcome 1, analysis 1]; Test type: Other — Concordance between 0.40 mercury and 0.5% elemental mercury in petrolatum; Kappa statistic = 0.67, 95% CI 2-sided [0.35 to 0.99]
Statistical Analysis 3: Comparison: Ammoniated Mercury; [analysis description as in outcome 1, analysis 1]; Test type: Other — Concordance between 0.36 mg/cm2 mercury and 1.0% ammoniated mercury in petrolatum; Kappa statistic = 0.46, 95% CI 2-sided [0.15 to 0.76]
Statistical Analysis 4: Comparison: Ammoniated Mercury; [analysis description as in outcome 1, analysis 1]; Test type: Other — Concordance between 0.36 mg/cm2 mercury and 0.5% elemental mercury in petrolatum; Kappa statistic = 0.57, 95% CI 2-sided [0.21 to 0.93]
Statistical Analysis 5: Comparison: Sodium Tetrachloropalladaate (Palladium); [analysis description as in outcome 1, analysis 1]; Test type: Other — Concordance between 0.10 mg/cm2 palladium and 3.0% sodium tetrachloropalladate in petrolatum; Kappa statistic = 0.48, 95% CI 2-sided [0.05 to 0.90]
Statistical Analysis 6: Comparison: Sodium Tetrachloropalladaate (Palladium); [analysis description as in outcome 1, analysis 1]; Test type: Other — Concordance between 0.10 mg/cm2 palladium and 1.0% palladium chloride in petrolatum; Kappa statistic = 0.39, 95% CI 2-sided [0.10 to 0.68]
Statistical Analysis 7: Comparison: Sodium Tetrachloropalladaate (Palladium); Concordance between 0.30 mg/cm2 palladium and 3.0% sodium tetrachloropalladate in petrolatum; Test type: Other; Kappa statistic = 0.83, 95% CI 2-sided [0.50 to 1.00]
Statistical Analysis 8: Comparison: Sodium Tetrachloropalladaate (Palladium); [analysis description as in outcome 1, analysis 1]; Test type: Other — Concordance between 0.30 mg/cm2 palladium and 1.0% palladium chloride in petrolatum; Kappa statistic = 0.19, 95% CI 2-sided [-0.02 to 0.39]
Statistical Analysis 9: Comparison: Sodium Tetrachloropalladaate (Palladium); [analysis description as in outcome 1, analysis 1]; Test type: Other — Concordance between 0.60 mg/cm2 palladium and 3.0% sodium tetrachloropalladate in petrolatum; Kappa statistic = 0.83, 95% CI 2-sided [0.50 to 1.00]
Statistical Analysis 10: Comparison: Sodium Tetrachloropalladaate (Palladium); [analysis description as in outcome 1, analysis 1]; Test type: Other; Concordance between 0.60 mg/cm2 palladium and 1.0 palladium chloride in petrolatum; Kappa statistic = 0.06, 95% CI 2-sided [-0.05 to 0.17]

2. Secondary Outcome: Number of Participants Who Exhibit Tape Irritation, Itching and Burning Resulting From Patch Test Panel Application.
Description: Tape irritation is graded on a 4 point scale: None (no tape irritation), Weak (faint to definite pink), Moderate (moderate erythema, definite redness) and Strong (severe erythema, very intense redness). Percentage of response will include weak, moderate and strong reactions.
  Itching and Burning are graded on a 4 point scale: None (no discomfort), Weak (minimal discomfort), Moderate (definite discomfort) and Strong (significantly bothersome, possible interference with sleep or daily activity). Percentage of response will include weak, moderate and strong responses.
Time Frame: Day 2: 48 hours after application
Measure: Count of Participants; unit: Participants
Arm/Group | Ammoniated Mercury | Aluminum Chloride and Aluminum Lactate | Sodium Tetrachloropalladaate (Palladium)
Number analyzed (Participants) | 21 | 13 | 21
Participants
  Tape Irritation: None | 17 | 9 | 21
  Tape Irritation: Weak | 4 | 2 | 0
  Tape Irritation: Moderate | 0 | 2 | 0
  Tape Irritation: Strong | 0 | 0 | 0
  Itching: None | 12 | 4 | 6
  Itching: Weak | 8 | 4 | 9
  Itching: Moderate | 1 | 2 | 5
  Itching: Strong | 0 | 3 | 1
  Burning: None | 20 | 9 | 19
  Burning: Weak | 1 | 3 | 1
  Burning: Moderate | 0 | 0 | 1
  Burning: Strong | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were reported beginning at the 2nd visit (day 2) through the end of the study, (day 19-23)
Description: Subjects were asked at each visit if they had any changes to their general health or use of concomitant medications
Groups:
- Ammoniated Mercury: Subjects will be patch tested with 4 experimental doses of ammoniated mercury, 0.013 mg/cm², 0.040 mg/cm², 0.12 mg/cm², and 0.36 mg/cm², a negative control and corresponding reference allergens, 1.0% ammoniated mercury in petrolatum and 0.5% elemental mercury in petrolatum. Patch tests will be worn for 48 hours.
  It was impossible to know which allergen dose was associated with a related adverse event
- Aluminum Chloride and Aluminum Lactate: Subjects will be patch tested with 4 experimental doses of aluminum chloride, 0.040 mg/cm², 0.12 mg/cm², 0.36 mg/cm² and 0.72 mg/cm², 4 experimental doses of aluminum lactate 0.047 mg/cm², 0.14 mg/cm², 0.42 mg/cm² and 0.84 mg/cm², a negative control and corresponding reference allergens, 2.0% aluminum chloride in petrolatum and 12.0% aluminum lactate in petrolatum. Patch tests will be worn for 48 hours.
  It was impossible to know which allergen dose was associated with a related adverse event
- Sodium Tetrachloropalladaate (Palladium): Subjects will be patch tested with 5 experimental doses of sodium tetrachloropalladate 0.011 mg/cm², 0.033 mg/cm², 0.10 mg/cm², 0.30 mg/cm² and 0.60 mg/cm², a negative control and corresponding reference allergens, 3.0% sodium tetrachloropalladate in petrolatum and 1.0% palladium chloride 1.0% in petrolatum. Patch tests will be worn for 48 hours.
  It was impossible to know which allergen dose was associated with a related adverse event
Arm/Group | Ammoniated Mercury | Aluminum Chloride and Aluminum Lactate | Sodium Tetrachloropalladaate (Palladium)
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/13 | 0/22
Serious Adverse Events (participants affected / at risk) | 1/21 | 0/13 | 0/22
Other Adverse Events (participants affected / at risk) | 6/21 | 3/13 | 9/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ammoniated Mercury (N=21) | Aluminum Chloride and Aluminum Lactate (N=13) | Sodium Tetrachloropalladaate (Palladium) (N=22)
Shock hypoglycemic (Metabolism and nutrition disorders) | 1 (1) | NA | NA — Emergency services called for insulin shock. Subject administered sugar infusion and Novorapid. Event resolved same evening. Investigator considered event serious but as it did not meet the criteria for an SAE it was not reported as such.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ammoniated Mercury (N=21) | Aluminum Chloride and Aluminum Lactate (N=13) | Sodium Tetrachloropalladaate (Palladium) (N=22)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (11) | 0 | 0 — Muscle pain, left side of torso
Blister (Skin and subcutaneous tissue disorders) | 1 (11) | 0 | 0 — Vesicles in nose
Blister (Skin and subcutaneous tissue disorders) | 1 (11) | 0 | 0 — Vesicles in mouth
Blister (Skin and subcutaneous tissue disorders) | 1 (11) | 0 | 0 — Vesicles on foot
Blister (Skin and subcutaneous tissue disorders) | 1 (11) | 0 | 0 — Vesicles on fingers
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 (5) | 0 — Acne-like lesions on posterior aspect of trunk
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 (11) — Allergic reaction on upper posterior aspect of trunk
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 (5) | 0 — Bilateral upper arm pruritus
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 (5) | 0 — Eczema in both axillae
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (11) — Erythematous scaling on no. 3 fingers, both hands
Pyrexia (General disorders) | 1 (11) | 0 | 0 — Fever
Headache (Nervous system disorders) | 0 | 0 | 1 (11) — Headache
Herpes Zoster (Infections and infestations) | 0 | 0 | 1 (11) — Herpes Zoster
Herpes (Infections and infestations) | 1 (11) | 0 | 0 — Herpes zoster on the back
Application site pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 (11) — Itching on the back patch test sites- left side
Lichenification (Skin and subcutaneous tissue disorders) | 1 (11) | 0 | 0 — Oral lichenoid lesions, left side
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (11) — Pain in shoulder
Application site papules (Skin and subcutaneous tissue disorders) | 0 | 1 (5) | 0 — Papules on upper posterior aspect of trunk
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (11) — Pruritus on back
Application site pruritus (Skin and subcutaneous tissue disorders) | 1 (11) | 0 | 1 (11) — Pruritus on the back at the test area
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 (11) — Pruritus on left side of back
Complex regional pain (Nervous system disorders) | 1 (11) | 0 | 0 — Upper back causalgia
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 (5) | 0 — Pruritus on upper posterior aspect of trunk
Upper respiratory tract infection (Infections and infestations) | 1 (11) | 0 | 0 — Upper respiratory tract infection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No